CLINICAL TRIAL: NCT04218110
Title: Preoperative Skin Preparation Study Following ASTM E1173 Methods to Evaluate the Antimicrobial Capabilities of Four Test Substances
Brief Title: Preoperative Skin Preparation Study to Evaluate the Antimicrobial Capabilities of Four Test Substances
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Professional Disposables International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ER19/232
Record Dates: First submitted 2019-12-30; First posted 2020-01-06 (Actual); Results first posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Surgical Site Infection
Keywords: Preventative
MeSH Terms: conditions — Surgical Wound Infection | interventions — 2-Propanol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Samples are blinded to the Microbiology group, participant, sponsor (1 of 2) and statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Project X 26ml (Experimental): 3.15% w/v CHG (chlorhexidine gluconate) /70% v/v IPA (isopropyl alcohol) contained within a saturated at use applicator. 26ml volume. Single use.
  Interventions: Drug: Isopropyl alcohol & Chlorhexidine Gluconate Antiseptic
- Project X 10.5ml (Experimental): 3.15% w/v CHG (chlorhexidine gluconate) /70% v/v IPA (isopropyl alcohol) contained within a saturated at use applicator. 10.5ml volume. Single use.
  Interventions: Drug: Isopropyl alcohol & Chlorhexidine Gluconate Antiseptic
- Project X 5.1ml (Experimental): 3.15% w/v CHG (chlorhexidine gluconate) /70% v/v IPA (isopropyl alcohol) contained within a saturated at use applicator. 10.5ml volume. Single use.
  Interventions: Drug: Isopropyl alcohol & Chlorhexidine Gluconate Antiseptic
- Prevantics Maxi Swabstick (Active Comparator): 3.15% w/v CHG (chlorhexidine gluconate) /70% v/v IPA (isopropyl alcohol) contained within pre-saturated applicator. 5.1ml volume. Single use.
  Interventions: Drug: Prevantics 3.15 % / 70 % Swabstick

INTERVENTIONS:
Drug: Isopropyl alcohol & Chlorhexidine Gluconate Antiseptic — Application of antiseptic drug to the inguinal area of the subjects
  Other Names: Project X 26ml
  Arms: Project X 26ml
Drug: Isopropyl alcohol & Chlorhexidine Gluconate Antiseptic — Application of antiseptic drug to the inguinal area of the subjects
  Other Names: Project X 10.5ml
  Arms: Project X 10.5ml
Drug: Isopropyl alcohol & Chlorhexidine Gluconate Antiseptic — Application of antiseptic drug to the inguinal area of the subjects
  Other Names: Project X 5.1ml
  Arms: Project X 5.1ml
Drug: Prevantics 3.15 % / 70 % Swabstick — Application of antiseptic drug to the inguinal area of the subjects
  Other Names: Prevantics Maxi Swabstick
  Arms: Prevantics Maxi Swabstick

SUMMARY:
Comparative study of antimicrobial effectiveness evaluation of of 26ml Project X, 10.5ml Project X, 5.1ml Project X and Prevantics Maxi swabstick following ASTM E1173 - Standard test method for evaluation of preoperative, precatheterization or preinjection skin preparations.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 18 years of age and of any race
2. In good general health
3. Read, understand and sign the Informed Consent Form (ICF)
4. If female of child-bearing potential, are willing to use an acceptable method of contraception to prevent pregnancy (i.e. oral contraceptive, intra-uterine device, diaphragm, condom, abstinence, bilateral tubal ligation, or are in a monogamous relationship with a partner who has had a vasectomy)
5. Female subjects of child-bearing potential, must have a negative Urine Pregnancy Test (UPT) on Treatment Day prior to any applications of the study products

Exclusion Criteria:

1. Exposure of test sites to antimicrobial agents, medicated soaps, medicated shampoos, or medicated lotions, use of biocide-treated pools or hot tubs, use of tanning beds, or sunbathing during the 14-day washout conditioning period and during the test period
2. Exposure of the test sites to strong detergents, solvents, or other irritants during the 14-day washout conditioning period and during the test period
3. Wear fabric softener, bug repellent or UV-treated clothing during the 14-day washout conditioning period and during the test period
4. Receive an irritation score of 1 (any redness, swelling, rash, or dryness present at any treatment area) for any individual skin condition prior to the Treatment Day baseline sample collection
5. Use of systemic or topical antibiotic medications, steroid medications (other than for hormonal contraception or post-menopausal reasons), or any other product known to affect the normal microbial flora of the skin during the 14-day washout conditioning period and during the test period
6. Known allergies or sensitivities to vinyl, latex (rubber), alcohols, metals, inks, or tape adhesives, or to common antibacterial agents found in soaps, lotions, or ointments, particularly isopropyl alcohol or chlorhexidine gluconate
7. A medical diagnosis of a physical condition, such as a current or recent severe illness, asthma, diabetes, hepatitis, an organ transplant, mitral valve prolapses, congenital heart disease, internal prostheses, or any immunocompromised conditions such as AIDS (or HIV positive)
8. Pregnancy, plans to become pregnant within the washout and test periods of the study, or nursing a child
9. Any tattoos or scars within 2" (5.08 cm) of the test sites
10. Dermatoses, cuts, lesions, active skin rashes, or breaks or other skin disorders within 6" on or around the test sites
11. A currently active skin disease or inflammatory skin condition (for example, contact dermatitis) anywhere on the body that, in the opinion of the Consulting Physician or PI, would compromise subject safety or study integrity
12. Showering, bathing, or swimming within the 72-hour period prior to sampling for Treatment Day, and throughout the test period
13. Participation in another clinical study in the past 30 days or current participation in another clinical study at time of signing informed consent
14. Any medical condition or use of any medications that, in the opinion of the PI, should preclude participation
15. Unwillingness to fulfill the performance requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rozalia Olsavszky, MD, Principal Investigator — EUROFINS EVIC PRODUCT TESTING ROMANIA S.R.L
Locations (1):
- Eurofins EVIC, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 328 individual subjects were consented, screened, treated and completed the study. Each subject is able to receive 2 test products (1 on each side of their body).
Groups:
- Project X 26ml: 3.15% w/v CHG (chlorhexidine gluconate)/70% v/v IPA (isopropyl alcohol) contained within a saturated at use applicator. 26ml volume. Single use.
  Isopropyl alcohol & Chlorhexidine Gluconate Antiseptic: Application of antiseptic drug to the inguinal area of the subjects
- Project X 10.5ml; Project X 5.1ml: 3.15% w/v CHG (chlorhexidine gluconate)/70% v/v IPA (isopropyl alcohol) contained within a saturated at use applicator. 10.5ml volume. Single use.
  Isopropyl alcohol & Chlorhexidine Gluconate Antiseptic: Application of antiseptic drug to the inguinal area of the subjects
- Prevantics Maxi Swabstick: 3.15% w/v CHG (chlorhexidine gluconate)/70% v/v IPA (isopropyl alcohol) contained within pre-saturated applicator. 5.1ml volume. Single use.
  Prevantics 3.15 % / 70 % Swabstick: Application of antiseptic drug to the inguinal area of the subjects
Period: Overall Study
Arm/Group | Project X 26ml | Project X 10.5ml | Project X 5.1ml | Prevantics Maxi Swabstick
Started | 82 | 81 | 83 | 83
Received Treatment | 82 | 81 | 83 | 82
Completed | 82 | 81 | 83 | 82
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Participant data is based on the Intent to Treat (ITT) data set.
Groups:
- Project X 26ml: 3.15% w/v CHG/70% v/v IPA contained within a saturated at use applicator. 26ml volume. Single use.
  Isopropyl alcohol & Chlorhexidine Gluconate Antiseptic: Application of antiseptic drug to the inguinal area of the subjects
- Project X 10.5ml; Project X 5.1ml: 3.15% w/v CHG/70% v/v IPA contained within a saturated at use applicator. 10.5ml volume. Single use.
  Isopropyl alcohol & Chlorhexidine Gluconate Antiseptic: Application of antiseptic drug to the inguinal area of the subjects
- Prevantics Maxi Swabstick: 3.15% w/v CHG/70% v/v IPA contained within pre-saturated applicator. 5.1ml volume. Single use.
  Prevantics 3.15 % / 70 % Swabstick: Application of antiseptic drug to the inguinal area of the subjects
- Total: Total of all reporting groups
Arm/Group | Project X 26ml | Project X 10.5ml | Project X 5.1ml | Prevantics Maxi Swabstick | Total
Number analyzed (Participants) | 82 | 81 | 83 | 83 | 329
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.76 (9.54) | 54.39 (11.70) | 54.48 (10.99) | 55.06 (10.23) | 54.67 (10.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 74 | 71 | 72 | 294
  Male | 5 | 7 | 12 | 11 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 82 | 81 | 83 | 83 | 329
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 81 | 81 | 83 | 82 | 327
  American Indian/Alaska Native | 0 | 0 | 0 | 0 | 0
  Black/African American | 1 | 0 | 0 | 1 | 2
  Asian | 0 | 0 | 0 | 0 | 0
  Subject Refused to Disclose | 0 | 0 | 0 | 0 | 0
  Other/Combination of 2 or more races (specify) | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Romania | 82 | 81 | 83 | 83 | 329
Weight [Mean (Standard Deviation); unit: kg] | 74.49 (13.98) | 73.37 (13.84) | 75.04 (16.11) | 74.98 (15.06) | 74.47 (14.77)
Height [Mean (Standard Deviation); unit: cm] | 163.03 (6.56) | 163.54 (7.84) | 164.65 (8.13) | 164.15 (7.85) | 163.84 (7.63)

OUTCOME MEASURES:

1. Primary Outcome: Change in Bacterial Microflora in the Inguinal Area
Description: Bacterial microflora (log10) will be measured via cup scrub method following the administration of the intervention
Time Frame: 10 minutes
Population: The Overall Number of Participants Analyzed represents the modified intent to treat (mITT) dataset where the Participant Flow represents the intent to treat (ITT) dataset. Additionally, each subject is able to receive 2 test products (1 on each side of their body).
Measure: Mean (Standard Deviation); unit: log10 CFU
Units Other Than Participants: evaluable sites
Arm/Group | Project X 26ml | Project X 10.5ml | Project X 5.1ml | Prevantics Maxi Swabstick
Number analyzed (Participants) | 44 | 42 | 47 | 45
Number analyzed (evaluable sites) | 88 | 84 | 93 | 89
log10 CFU | -3.86 (1.58) | -4.34 (1.48) | -3.65 (1.36) | -3.80 (1.42)

2. Secondary Outcome: Change in Bacterial Microflora in the Inguinal Area
Description: Bacterial microflora (log10) will be measured via cup scrub method following the administration of the intervention
Time Frame: 30 seconds
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 CFU
Units Other Than Participants: evaluable sites
Arm/Group | Project X 26ml | Project X 10.5ml | Project X 5.1ml | Prevantics Maxi Swabstick
Number analyzed (Participants) | 44 | 42 | 47 | 45
Number analyzed (evaluable sites) | 88 | 84 | 93 | 89
log10 CFU | -3.86 (1.55) | -3.76 (1.36) | -3.70 (1.58) | -3.76 (1.48)

ADVERSE EVENTS:
Time Frame: 1.5 months
Arm/Group | Project X 26ml | Project X 10.5ml | Project X 5.1ml | Prevantics Maxi Swabstick
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/81 | 0/83 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/81 | 0/83 | 0/82
Other Adverse Events (participants affected / at risk) | 0/82 | 0/81 | 0/83 | 0/82
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Project X 26ml (N=82) | Project X 10.5ml (N=81) | Project X 5.1ml (N=83) | Prevantics Maxi Swabstick (N=82)
Adverse Event (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unexpected, non-serious adverse event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-29): https://cdn.clinicaltrials.gov/large-docs/10/NCT04218110/Prot_SAP_000.pdf